## 16.1.9 Documentation of Statistical Methods

Paion UK Ltd., Statistical Analysis Plan, Final Version 1.0, dated 09-Jun-2017

Paion UK Ltd., Statistical Analysis Plan Tables Figures, Listing TOCs, Final Version 1.0, dated 09-Jun-2017



## STATISTICAL ANALYSIS PLAN

Title: A Phase III Study Evaluating the Efficacy and Safety of

Remimazolam (CNS 7056) Compared to Placebo and Midazolam in Patients Undergoing Bronchoscopy

**Protocol Number:** CNS7056-008

**Compound:** Remimazolam

Phase: III

**Sponsor:** PAION UK Ltd

**Author:** 

Date: 09 June 2017

Version: Final 1.0



Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

#### STATISTICAL ANALYSIS PLAN APPROVALS



# **Table of Contents**

| 1 | <b>OVERVIEV</b> | W | 10 |
|---|---|---|---|
| 2 | STUDY OF | BJECTIVES AND ENDPOINTS | 11 |
| | 2.1 | Primary Objective | 11 |
| | 2.2 | Secondary Objectives | 11 |
| | 2.3 | Safety and Efficacy Endpoints | 11 |
| | 2.3.1 | Efficacy Endpoints | 11 |
| | 2.3.1.1 | Primary Efficacy Endpoints | 11 |
| | 2.3.1.2 | Secondary Efficacy Endpoints | 11 |
| | 2.3.2 | Safety Endpoints | 12 |
| | 2.3.3 | | |
| 3 | OVERALL | STUDY DESIGN AND PLAN | 14 |
| | 3.1 | Study Population | 15 |
| | 3.2 | Method of Assigning Patients to Treatment Groups | 15 |
| | 3.3 | Treatment Blinding | 16 |
| | 3.4 | Schedule of Assessments | 16 |
| | 3.5 | Sample Size Calculation | 16 |
| 4 | ANALYSIS | S AND REPORTING | 18 |
| | 4.1 | Software and general statistical methods | 18 |
| | 4.2 | Interim Analyses and Data Monitoring | 18 |
| | 4.3 | Final Analysis | 18 |
| 5 | ANALYSIS | S POPULATIONS | 19 |
| 6 | GENERAL | ISSUES FOR STATISTICAL ANALYSIS | 20 |
| | 6.1 | General Statistical Methodology | 20 |
| | 6.1.1 | Adjustments for Multiple Comparisons | 20 |
| | 6.1.2 | Methods for Dropouts or Missing Data | 20 |
| | 6.1.3 | Pooling of Centers | 20 |
| | 6.1.4 | Analysis Visit Windows | 20 |
| | 6.1.5 | Data Handling Conventions | 20 |
| | 6.1.5.1 | Baseline Definitions | 20 |
| | 6.1.5.2 | Start Date, End Date of Study Treatment, and Study Day | 21 |

| | 6.1.5.3 | Early Termination (ET) Visit | 21 |
|---|---|---|---|
| | 6.1.5.4 | Unscheduled Visits | 21 |
| | 6.1.5.5 | Incomplete Date and Time Imputation for Adverse Events and Concomitant Medications | 21 |
| | 6.1.6 | By Patient Data Listings | 23 |
| | 6.2 | Derived and Computed Variables | 23 |
| 7 | STUDY PAT | TIENTS AND DEMOGRAPHICS | 28 |
| | 7.1 | Disposition of Patients and Withdrawals | 28 |
| | 7.2 | Protocol Deviations. | 28 |
| | 7.3 | Demographics and Baseline Characteristics | 28 |
| | 7.4 | Medical History | 28 |
| 8 | EFFICACY A | ANALYSIS | 29 |
| | 8.1 | Primary Efficacy | 29 |
| | 8.1.1 | Primary Efficacy Endpoint | 29 |
| | 8.1.2 | Primary Analysis | 29 |
| | 8.1.3 | | |
| | 8.2 | Secondary Efficacy | 30 |
| 9 | SAFETY AN | ID TOLERABILITY ANALYSIS | 33 |
| | 9.1 | Adverse Events | 33 |
| | 9.1.1 | | |
| | 9.1.5.1 | | |
| | 9.1.2<br>Associated w | Adverse Events Related to Effects Seen with Medications Known to ith Abuse | |
| | 9.2 | Clinical Laboratory Tests | 35 |
| | 9.3 | Vital Signs, Pulse Oximetry | 36 |
| | 9.3.1 | Continuous Monitoring | 36 |
| | 9.3.2 | Continuous Monitoring – Exploratory Analyses | 37 |
| | 9.4 | Electrocardiograms | 37 |
| | 9.4.1 | 12-Lead ECG | 37 |
| | 9.4.2 | 3-Lead ECG | 37 |
| | 9.5 | Physical Examinations | 37 |
| | 9.6 | | |
| | 9.7 | Prior and Concomitant Medications | 38 |

| | 9.7.1 | Prior and Concomitant Medications | 38 |
|---|---|---|---|
| | 9.7.2 | Rescue Sedative Medications | 38 |
| 9 | .8 | | |
| 10 | CHANGE | ES TO PLANNED ANALYSES | 40 |
| 11 | REFERENCES4 | | |
| 12 | ATTACH | IMENTS | 42 |
| | APPEN | NDIX A: Details of AEs with a Respiratory or Cardiovascular Focus | 43 |
| | APPEN | NDIX B: Diseases of Interest for Drug-Disease Interaction Analysis | 55 |

09 June 2017

# LIST OF ABBREVIATIONS

| χ²chi-squaredAEAdverse eventAESIAdverse event of special interestANOVAAnalysis of varianceASA-PSAmerican Society of Anesthesiologists-Physical StatusATCAnatomical Therapeutic ClassAUCArea under the curveBPBlood pressurebpmBeats per minuteBMIBody mass indexCMHCochran-Mantel-HaenszelCNS 7056BCNS 7056 besylatecmCentimeter(s) | Definition |
|---|---|
| AESI Adverse event of special interest ANOVA Analysis of variance ASA-PS American Society of Anesthesiologists-Physical Status ATC Anatomical Therapeutic Class AUC Area under the curve BP Blood pressure bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | |
| ANOVA Analysis of variance ASA-PS American Society of Anesthesiologists-Physical Status ATC Anatomical Therapeutic Class AUC Area under the curve BP Blood pressure bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | |
| ASA-PS American Society of Anesthesiologists-Physical Status ATC Anatomical Therapeutic Class AUC Area under the curve BP Blood pressure bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | Adverse event of special interest |
| ATC Anatomical Therapeutic Class AUC Area under the curve BP Blood pressure bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | Analysis of variance |
| AUC Area under the curve BP Blood pressure bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | |
| BP Blood pressure bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | Anatomical Therapeutic Class |
| bpm Beats per minute BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | |
| BMI Body mass index CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | |
| CMH Cochran-Mantel-Haenszel CNS 7056B CNS 7056 besylate | |
| CNS 7056B CNS 7056 besylate | |
| · | |
| cm Centimeter(s) | |
| CM Concomitant medication | |
| CRF Case report form | |
| CS Clinically significant | |
| CSR Clinical study report | |
| CTA Clinical Trial Agreement | |
| ECG Electrocardiogram | |
| EMA European Medicines Agency | |
| ET Early termination | |

| Protocol | l CNS7056-008 | ' Statistical | l Analysis Plan |
|----------|---------------|---------------|-----------------|
|----------|---------------|---------------|-----------------|

09 June 2017

| Abbreviation | Definition |
|--------------|----------------------------------------------------------|
| FDA | Food and Drug Administration |
| GCP | Good clinical practice |
| h | Hour(s) |
| ICH | International Conference on Harmonization |
| IMP | Investigational Medicinal Product |
| ITT | Intent-to-treat |
| IWRS | Interactive web response system |
| kg | Kilogram(s) |
| LOCF | Last observation carried forward |
| LS | Least squares |
| max | maximum |
| μg | Microgram |
| mg | Milligram |
| min | Minute(s) |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-treat |
| MOAA/S | Modified Observer's Assessment of Alertness and Sedation |
| MON | Month |
| NDA | New Drug Application |
| NRS | Numeric rating scale |
| PP | Per protocol |

| D 1 010707070000000000000000000000000000 | 00 7 2017 |
|------------------------------------------------|--------------|
| Protocol CNS7056-008 Statistical Analysis Plan | 09 June 2017 |

| Abbreviation | Definition |
|---|---|
| QTc | Corrected QT interval |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SMQ | Standardised MedDRA query |
| SOC | System organ class |
| $\mathrm{SpO}_2$ | Peripheral blood oxygen saturation (measured by pulse oximetry) |
| TEAE | Treatment-emergent adverse event |
| TRTM | Month of start of study treatment |
| TRTY | Year of start of study treatment |
| USA | United States of America |
| yr | Year |
| YYYY | Year |
| WHO-DD | World Health Organization – Drug Dictionary |

#### 1 OVERVIEW

This document presents a detailed statistical analysis plan for the available data from Paion's protocol CNS7056-008, Amendment 5.0, dated 3 March 2016 (A Phase III Study Evaluating the Efficacy and Safety of Remimazolam (CNS 7056) Compared to Placebo and Midazolam in Patients Undergoing Bronchoscopy).

Reference materials for this statistical plan include Protocol CNS7056-008 version 1.0 Amendment 5.0, dated 03-Mar-2016 and the accompanying SDTM and ADaM specification documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this statistical analysis plan (SAP) unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials [1]. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association [2] and the Royal Statistical Society [3], for statistical practice.

All planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analysis not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc, or unplanned, exploratory analyses performed will be clearly identified as such in the final CSR.

#### 2 STUDY OBJECTIVES AND ENDPOINTS

## 2.1 Primary Objective

The objective is to establish the superiority of remimazolam compared to placebo in inducing and maintaining suitable sedation levels for patients undergoing bronchoscopy and to assess data from an additional open-label midazolam group in combination with fentanyl as determined by sedation success.

## 2.2 Secondary Objectives

Secondary objectives include assessing time to event endpoints (as described in detail under Section 2.3.1.2 Secondary Efficacy Endpoints).

## 2.3 Safety and Efficacy Endpoints

## 2.3.1 Efficacy Endpoints

#### 2.3.1.1 Primary Efficacy Endpoints

The primary efficacy endpoint is to assess the success of sedation of the bronchoscopy procedure. This composite endpoint will be determined for remimazolam and placebo by the following criteria:

- Completion of the bronchoscopy procedure, AND
- No requirement for a rescue sedative medication, AND
- No requirement for more than 5 doses of study medication within any 15 minute window in the blinded arms (remimazolam/placebo) or no requirement for more than 3 doses within any 12 minute window in the open-label midazolam arm.

#### 2.3.1.2 Secondary Efficacy Endpoints

Secondary efficacy endpoints are:

- 1. The **time to start of procedure** after administration of the first dose of study medication.
- 2.
- 3. The **time to ready for discharge** (defined as ability to walk unassisted) after the end of bronchoscopy procedure (bronchoscope out).
- 4. The **time to ready for discharge** after the last injection of study drug.

- 5. The **times to fully alert** (time to first of three consecutive Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scores of 5) after the end of bronchoscopy procedure (bronchoscope out)).
- 6. The **times to fully alert** (time to first of three consecutive MOAA/S scores of 5) after the last injection of study drug).



#### 2.3.2 Safety Endpoints

Safety endpoints include:

- 1. Adverse events (AEs)
- 2. Clinical laboratory test results
- 3. Vital signs (supine heart rate, systolic and diastolic blood pressure (BP), calculated mean arterial pressure, respiration rate, temperature)
- 4. Pulse oximetry measurements (presented by patient for pre-defined time points, and as oxygen saturation over time (AUC))
- 5. Electrocardiogram (ECG) findings
- 6. Physical examination findings
- 7.
- 8.



10. The safety of multiple doses (initial dose and additional top-up doses) of remimazolam including oxygen saturation and no need for mechanical ventilation following administration of a standard dose of fentanyl.



#### 3 OVERALL STUDY DESIGN AND PLAN

This study is a prospective, randomized, placebo and active controlled, multi-center, parallel group study comparing remimazolam to placebo in a double-blind manner, with an additional open-label midazolam arm, in patients undergoing bronchoscopy. 420 patients will be randomized into one of three possible study groups: placebo (n=60), midazolam (n=60), and remimazolam (n=300).

All patients will receive 0.9% NaCl solution up to 1000 mL drip starting prior to the procedure, if their fluid status allows. All patients will receive 25-50 µg of fentanyl immediately prior to the administration of study medication (with suitable dose reductions at the investigator's discretion for elderly and debilitated patients). All infused fluid volumes will be recorded throughout the procedure. The administration of supplemental oxygen will be started shortly before the procedure and will be continued at a rate of 4 L/min until the patient is fully alert (first of three consecutive MOAA/S scores of 5).

#### Blinded arms:

Patients will be randomized to manually receive an initial single intravenous (iv) dose over one minute of remimazolam 5.0 mg or an equal volume of placebo in a blinded manner and bronchoscopy will start when adequate sedation (MOAA/S  $\leq$ 3) has been achieved.

Sedation may be maintained by injection of further doses of remimazolam 2.5 mg or placebo in the same volume not earlier than two minutes apart after assessment of the sedative effect. The overall number of remimazolam/placebo doses is not limited as long as not more than 5 doses are administered in any 15 minute window. Should **five doses within 15 minutes** not be sufficient to obtain adequate sedation for the bronchoscopy, this is defined as a treatment failure.

#### Open-label arm:

In the open-label midazolam arm, healthy adults <60 years will receive 1.75 mg of midazolam as an initial dose over two minutes. Adults  $\ge60$  years, debilitated or chronically ill patients will receive 1.0 mg midazolam as an initial dose over two minutes. Sedation can be maintained by further doses of 1.0 mg in healthy adults <60 years; in the case of adults  $\ge60$  years, debilitated or chronically ill patients, the dose will be 0.5 mg. These subsequent doses should always be titrated slowly and administered over at least two minutes. At least two additional or more minutes should be allowed to fully evaluate the sedative effect. The overall number of midazolam doses is not limited as long as not more than three doses are administered in any 12 minute window. Should **three doses within any 12 minute** window not be sufficient to obtain adequate sedation for the bronchoscopy, this is to be considered a treatment failure.

After determination of treatment failure, midazolam is defined as the only rescue sedative medication in such cases in order to perform or finalize the bronchoscopy.

If the pain is not adequately controlled by the initial dose of 25-50  $\mu$ g fentanyl (with suitable dose reductions at the investigator's discretion for elderly and debilitated patients), further top up doses of fentanyl of 25  $\mu$ g q 5-10 minutes are allowed until adequate analgesia is achieved or the maximum dose of 200  $\mu$ g per procedure has been reached. It is of note, that fentanyl is strictly to be applied for pain control only.

## 3.1 Study Population

This is a study in patients undergoing a bronchoscopy for diagnostic or therapeutic purposes (e.g. biopsies, lavage, brushings, and foreign body extraction). A total of 420 patients will be randomized, of which 300 will receive remimazolam, 60 will receive placebo (0.9% NaCl) in a blinded fashion, and 60 patients will receive midazolam open label.

## 3.2 Method of Assigning Patients to Treatment Groups

Before dosing, patients will be randomly assigned in a 30:6:6 ratio to remimazolam, placebo or open-label midazolam. The randomization schedule will be computer-generated using a permuted block algorithm and will randomly allocate study drug to randomization numbers. The randomization numbers will be assigned sequentially as patients are entered into the study. The study site will not be stratified in the randomization schedule. Although the amount of chronic use of opioids and/or benzodiazepines will be known in advance, it is difficult to be able to stratify the randomization for amount of these drugs from a practical perspective.

Randomization will be stratified by age group. The aim is to have at least 100 patients on remimazolam aged  $\geq$  65 years (at least 30 of these aged  $\geq$  75 years or older) across the three late stage clinical trials (CNS7056-006, CNS7056-008, and CNS7056-015). The CNS7056-008 study will be included as part of an integrated analysis plan where age group will be assessed as above.

On Study Day 1, after confirming that a patient still meets entry criteria, study personnel will inform the pharmacist that the patient qualifies for randomization. The unblinded pharmacist will call the central interactive web response system (IWRS) and enter the requested information. The IWRS will then assign the next randomization number in the sequence and inform the pharmacist of the study treatment assignment. Thereafter, the pharmacist will dispense the corresponding treatment.

| Group | Trial medication | Initial dose + Top up dose |
|---|---|---|
| Group 1 (N = 60) | Placebo | Volume to match group 2 |
| Group 2 (N = 300) Remimazolam $5.0 \text{ mg} + 2.5 \text{ mg}$ | | 5.0 mg + 2.5 mg |
| Group 3 (N = 60) Midazolam $1.75 \text{ mg} + 1.0 \text{ mg}^* \text{ or } 1.0 \text{ mg} + 0.5 \text{ mg}^8$ | | 1.75 mg + 1.0 mg* or 1.0 mg + 0.5 mg <sup>§</sup> |
| *Healthy adults <60 years; §adults ≥60 years, debilitated or chronically ill patients. | | |

## 3.3 Treatment Blinding

The study will be conducted as a randomized, double-blind study with respect to remimazolam and placebo. The midazolam arm will be open-label. The identity of the blinded study drugs (remimazolam or placebo) will not be revealed to study management or to anyone at the study site except for the pharmacist, the pharmacy staff and unblinded monitor until the study is completed. This exemption also applies to the data monitoring committee (DMC) members. The pharmacist and staff will not participate in other study procedures. Patients will be blinded to treatment.

#### 3.4 Schedule of Assessments

The maximum study duration for any patient will be up to 28 days. The patients will be screened within 21 days prior to the bronchoscopy. A follow-up phone call will be performed on Day 4 (+3/-1 days) following the bronchoscopy.

<u>Screening (Day -21 to Day 1)</u>: Patients will sign informed consent and undergo procedures to determine eligibility.

Day of Bronchoscopy (Day 1): After the completion of screening procedures patients will be randomly assigned to the remimazolam, placebo or midazolam group. All patients will receive 25-50 μg of fentanyl immediately prior to the administration of study medication (with suitable dose reductions at the investigator's discretion for elderly and debilitated patients). Following completion of the bronchoscopy procedure, the patients will be discharged at the discretion of the investigator and complete the assessments after reaching fully alert status. Assessment of "time back to normal" in the patient's subjective view will be collected via telephone contact by study nurse on Day 2.

<u>Follow-up (Day 4 [+3/-1 days])</u>: The site will telephone the patient for safety assessments. Study participation is considered complete after all Day 4 assessments have been performed and all AEs have been followed-up until they resolve or become stable, or until they can be explained by another known cause(s).

In case there has been any indication for the onset of a new AE since discharge, patients should come back to the site immediately (preferably the same day) to perform further assessments (e.g.clinically laboratory tests, 12 lead ECG, left to the discretion of the investigator).



Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017



A total of 420 patients will be randomized, 300 to receive remimazolam, 60 to receive open-label midazolam, and 60 to receive placebo.

#### 4 ANALYSIS AND REPORTING

## 4.1 Software and general statistical methods

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.3 or higher) for Windows. If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

All measured variables and derived parameters will be listed individually and, if appropriate, tabulated by descriptive statistics.

For continuous variables, summary statistics including number of patients with data, mean, standard deviation (SD), median, minimum and maximum will be provided. For categorical variables, the number of patients and percentage for each category will be presented.

A blinded data review will be performed before the database is locked and the study groups are unblinded.

Study medication is defined as any of fentanyl or remimazolam, placebo or midazolam administered for the initial dosing or top-up doses.

Randomized study medication is defined as the Investigational Medicinal Product IMP (remimazolam, placebo or midazolam). The start of the initial dose of randomized study drug infusion will be considered Time 0 (t=0).

## 4.2 Interim Analyses and Data Monitoring

No interim analyses are planned for this study.

# 4.3 Final Analysis

All final, planned, analyses identified in the protocol and in this SAP will be performed only after the last patient has completed the last study visit and end of study assessments, all relevant study data have been processed and integrated into the analysis data base, and the clinical database has been locked and the randomization code has been unblinded. In addition, no database may be locked, randomization code unblinded, or analyses completed until this SAP has been approved.

All statistics and study results will be made available to Paion after database lock and before completion of the final CSR.



Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

#### 5 ANALYSIS POPULATIONS

Eight analysis populations are defined:

• The Safety Population will consist of all randomized patients who receive any amount of study drug and will be analyzed as treated.



- The Intent-to-treat analysis set (ITT) will include all patients who were randomized and will be analyzed as randomized.
- The Modified Intent-to-treat analysis set (mITT) will include all patients included in the ITT population who received at least one complete dose of randomised study medication. These will be analysed as randomized.
- The Per-Protocol analysis set (PP) will include all patients from the ITT analysis set who
  - received randomized treatment according to their randomization and the planned treatment schedule.
  - did not have any major protocol deviations

Protocol deviations to be considered are defined in the Protocol Deviation Guidance Plan.

Membership in the analysis populations will be determined before unblinding at the blinded data review meeting.



#### 6 GENERAL ISSUES FOR STATISTICAL ANALYSIS

## 6.1 General Statistical Methodology

#### 6.1.1 Adjustments for Multiple Comparisons

No adjustment for multiple testing is required for the primary endpoint as only one pairwise comparison will be performed between the remimazolam and placebo groups. Analyses of the remimazolam and placebo groups for all secondary parameters will be considered to be descriptive only as it is likely that most of the patients in the placebo group will have taken midazolam as rescue sedative medication. Therefore, these analyses will need to be interpreted with caution.

Comparison between the remimazolam and midazolam groups will be descriptive only, a 95% confidence interval of the difference will be presented but no further analysis will be performed.

#### 6.1.2 Methods for Dropouts or Missing Data

Incomplete dates and times for AEs and concomitant medications will be imputed as described in section 6.1.5.5 below.

Time to event variables will be censored as described in section 6.2 below if the event did not occur

#### 6.1.3 Pooling of Centers

The study will include data from all centers.

Centers who recruit fewer than 20 patients will be pooled into one "Other" center.

#### 6.1.4 Analysis Visit Windows

Analyses of all variables for this study will use the nominal visit or time point as collected in the case report form (CRF) and/or database.

#### 6.1.5 Data Handling Conventions

#### **6.1.5.1** Baseline Definitions

For all analyses, the baseline value is defined as the value recorded 'Within 5 hrs' or 'Within 15 minutes' before first dosing of study medication as shown in <u>Appendix B</u> Schedule of Assessments of the protocol. The most recent pre-dose value will be taken as baseline. Where a value is missing, the next previous value will be used.

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017

The date/time of the first dose (t=0) for the efficacy analyses is defined as the start date/time of first administration of randomized study medication.

Change from baseline will be defined as the Value – Baseline.

#### 6.1.5.2 Start Date, End Date of Study Treatment, and Study Day

The **start date of study treatment** is defined as the first date when study medication was taken (Day 1).

The **study day** for all assessments will be calculated using the start date of study treatment as the origin (Day 1):

```
study day = (date of assessment) - (start date of study treatment) + 1
```

For assessments/events with a date preceding the start date of study treatment, the following formula will be applied:

study day = (date of assessment) - (start date of study treatment)

#### 6.1.5.3 Early Termination (ET) Visit

Patients who discontinue from the study after randomization and before the Day 4 visit should be scheduled for an ET visit during which all assessments listed for the Day 4 visit will be performed.

#### 6.1.5.4 Unscheduled Visits

Data (such as laboratory tests and vital signs) collected at unscheduled visits will not be included in the analyses by scheduled visits, but may be used for baseline and for safety shift tables from baseline to most extreme value.

# 6.1.5.5 Incomplete Date and Time Imputation for Adverse Events and Concomitant Medications

For partial AE/concomitant medication (CM) start dates the imputation rules are described in the following table.

| Partial start date | | Date imputation |
|--------------------|-------------|--------------------------|
| YYYY missing | | No imputation |
| YYYY ≠ TRTY | MON missing | Imputed date = 01JANYYYY |

| Protocol CNS7056-008 Statistical Analysis Plan | 09 June 2017 |
|------------------------------------------------|--------------|
|------------------------------------------------|--------------|

| Partial start date | | Date imputation |
|---|---|---|
| YYYY ≠ TRTY | MON not missing,<br>DAY missing | Imputed date = 01MONYYYY |
| YYYY = TRTY | MON missing | Imputed date = start date of study treatment |
| YYYY = TRTY | MON < TRTM,<br>DAY missing | Imputed date = 01MONYYYY |
| YYYY = TRTY | MON ≥ TRTM,<br>DAY missing | Imputed date = max (01MONYYYY, start date of study treatment) |

YYYY=Year of AE/CM start date, MON=Month of AE/ CM start date, DAY=day of AE/ CM start date, TRTY=Year of start date of study treatment, TRTM=Month of start date of study treatment

For partial AE (or CM) end dates the imputation rules are defined as the following:

- If month or year of an AE (or medication) end date is missing, the AE (or medication) end date is set to the date of study completion/early termination.
- If day of an AE (or medication) end date is missing, but month and year of the AE (or medication) end date are not missing, the AE (or medication) end date is set to minimum of (end date of study treatment, last day of the month).

If an imputed AE (or CM) end date is earlier than the AE (or CM) start date, the AE (or CM) start date will be used as the imputed AE (or CM) end date.

After applying the rules above the following rules will be used to determine whether an AE is 'treatment emergent' or not and whether a medication is 'concomitant' or 'prior':

- If the start date is missing and the end date is either missing or on or after the start date of study treatment, then the AE (or medication) is considered to be treatment emergent (or concomitant).
- If the start time is missing and the start date is either on the same day as the start of study treatment or has been imputed as the same day as the start of study treatment, then the AE (or medication) is considered to be treatment emergent (or concomitant)
- If the start date is missing and the end date is before the start date of study treatment, then the AE (or medication) is considered to be not treatment emergent (or prior).
- If the start date is not missing and the end date is missing, then the medication is considered to be concomitant while the treatment emergent status is determined by the start date.

• If the start time in seconds is missing, then the seconds is replaced by a half-minute or 50 seconds.

## 6.1.6 By Patient Data Listings

All data available will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs, but will be included in the data listings.

## 6.2 Derived and Computed Variables

The following derived and computed variables have been initially identified as important for the analysis of the primary and secondary target variables. It is expected that additional variables will be required. The SAP will not be amended for additional variables that are not related to the primary target or key secondary target variables. Any additional derived or computed variables will be identified and documented in the SAS programs that create the analysis files. In all cases, incomplete dates will be completed for the analysis using a conservative/worst case solution.

| Variable<br>Name | Description | Valid<br>Values<br>(Ranges) | Computation Methods, Notes, or Equation(s) |
|---|---|---|---|
| SUCCESS | Overall Success<br>of the<br>Bronchoscopy<br>Procedure | 1 = Yes<br>0 = No | <ul> <li>SUCCESS = 1 if and only if all the following criteria are met:</li> <li>Completion of the bronchoscopy procedure</li> <li>No requirement for an alternative sedative medication</li> <li>No requirement for more than 5 doses of study medication (these 5 doses may include the initial dose) within any rolling 15 minute window in the double-blind arms or no requirement for more than 3 doses within any rolling 12 minute window in the open midazolam arm.</li> <li>Otherwise SUCCESS = 0</li> <li>The criterion of no more than 5 doses for a 15 minute window means that if any dose has a further 4 doses within the following 900 seconds inclusive, then SUCCESS = 0. The criterion for 3 doses within 12 minutes is defined similarly.</li> </ul> |
| T2START | Time to start of procedure | | T2START=1 + (start time of procedure) - (first dose of randomized study medication start time) in minutes For patients who do not start a procedure, this time will be censored at the time of dropout. |
| CENSOR2TS | Censor indicator for time to start of procedure | 1 = Yes<br>0 = No | If T2START was censored, CENSOR2TS = 1, else CENSOR2TS = 0. |

| Variable<br>Name | Description | Valid<br>Values<br>(Ranges) | Computation Methods, Notes, or Equation(s) |
|---|---|---|---|
| T2FAP | Time to Fully<br>Alert after the<br>end of the<br>procedure | | T2FAP = 1 + (time fully alert achieved) – (end time of procedure) in minutes, if patient reaches fully alert. Fully alert is defined as the first of three consecutive MOAA/S measurements of 5 after the end of the procedure. If a patient withdraws early, and/or does not reach Fully Alert at the end of the study, the patient's T2FAP will be censored using a patient's last MOAA/S assessment date. |
| CENSORAP | Censor Indicator<br>for Fully Alert<br>after the end of<br>the procedure | 1 = Yes<br>0 = No | If T2FAP was censored: CENSORAP=1; Else CENSORAP=0. |
| T2FAD | Time to Fully<br>Alert from the<br>end of the last<br>dose of study<br>drug or rescue<br>sedative drug | | T2FAD = 1+ (time fully alert achieved) – (end time of last dose of randomized study medication or rescue sedative medication) in minutes, if patient reaches fully alert. Fully Alert is defined as the first of three consecutive MOAA/S measurements of 5 after the start time of the last dose of study or rescue drug. If a patient withdraws early, and/or does not reach Fully Alert at the end of the study, the patient's T2FAD will be censored using a patient's last MOAA/S assessment. |
| CENSORAD | Censor Indicator<br>for Fully Alert<br>from the end of<br>the last dose of<br>study drug | 1 = Yes<br>0 = No | If T2FAD was censored: CENSORAD=1; Else CENSORAD=0. |

| Variable<br>Name | Description | Valid<br>Values<br>(Ranges) | Computation Methods, Notes, or Equation(s) |
|---|---|---|---|
| T2RDB | Time to Ready<br>for Discharge<br>from the end of<br>bronchoscopy<br>procedure | | T2RDB = 1 + (time ready for discharge) – (end time of bronchoscopy procedure) in minutes, if patient is ready for discharge. Ready for discharge is defined as ready to walk unassisted. If a patient withdraws early, and/or does not reach Ready for Discharge at the end of the study, the patient's T2RDB will be censored using the patient's last assessment. |
| CENSORDB | Censor Indicator<br>for Ready for<br>Discharge from<br>the end of<br>bronchoscopy<br>procedure | 1 = Yes<br>0 = No | If T2RDB was censored: CENSORDB = 1; Else CENSORDB = 0. |
| T2RDD | Time to Ready<br>for Discharge<br>from the end of<br>the last dose of<br>study drug. | | T2RDD = 1 + (time ready for discharge) – (end time of last dose of randomized study medication or rescue sedative medication) in minutes, if patient is ready for discharge. Ready for discharge is defined as ready to walk unassisted. If a patient withdraws early, and/or does not reach Ready for Discharge at the end of the study, the patient's T2RDD will be censored using the patient's last assessment. |
| CENSORDD | Censor Indicator<br>for Ready for<br>Discharge from<br>the end of the<br>last dose of<br>study drug. | 1 = Yes<br>0 = No | If T2RDD was censored: CENSORDB = 1; Else CENSORDB = 0. |

| Variable<br>Name | Description | Valid<br>Values<br>(Ranges) | Computation Methods, Notes, or Equation(s) |
|---|---|---|---|
| HRNADC | Lowest post-<br>dose value of<br>Heart Rate | | Lowest recorded post-dose value of Heart Rate in CRF on treatment day |
| RRNADC | Lowest post-<br>dose value of<br>Respiratory<br>Rate | | Lowest recorded post-dose value of Respiratory Rate in CRF on treatment day |

| Variable<br>Name | Description | Valid<br>Values<br>(Ranges) | Computation Methods, Notes, or Equation(s) |
|---|---|---|---|
| OXYNADC | Lowest post-<br>dose value of<br>SpO2 | | Lowest recorded post-dose value of SPO2 in CRF on treatment day |
| RRPEAK | Peak post-dose<br>value of<br>Respiratory<br>Rate | | Highest recorded post-dose value of Respiratory Rate in CRF on treatment day. |
| HRNADN | Lowest post-<br>dose value of<br>Heart Rate | | Lowest value of Heart Rate from Nellcor data on treatment day in the interval between the first dose of study medication and the time when the patient becomes fully alert |
| RRNADN | Lowest post-<br>dose value of<br>Respiratory<br>Rate | | Lowest value of Respiratory Rate from Nellcor data on treatment day in the interval between the first dose and the time when the patient becomes fully alert |
| OXYNADN | Lowest post-<br>dose value of<br>SpO2 | | Lowest value of SpO2 from Nellcor data on treatment day in the interval between the first dose and the time when the patient becomes fully alert |
| RRPEAKN | Peak post-dose<br>value of<br>Respiratory<br>Rate | | Highest value of Respiratory Rate from Nellcor data on treatment day in the interval between the first dose and the time when the patient becomes fully alert |

#### 7 STUDY PATIENTS AND DEMOGRAPHICS

## 7.1 Disposition of Patients and Withdrawals

The number of patients included in each analysis set (Safety, each Safety [Nellcor], ITT, mITT, PP) will be presented by treatment group and overall.

The number and percentage of patients who completed the study treatment period, who discontinued the study prior to the end of treatment and the reason for discontinuation, along with the number who completed the Follow-up Visit will be presented for each treatment group and overall, using the safety population.

All disposition summaries will also be presented by study center.

#### 7.2 Protocol Deviations

A list of protocol deviations that could affect the primary objective will be identified by the Clinical and Medical Monitors. This list will be finalized prior to database lock and unblinding of the study. The incidence of each protocol deviation will be presented for the ITT population.

## 7.3 Demographics and Baseline Characteristics

Demographics variables and baseline characteristics will be summarized for the safety population overall and by treatment group.

Demographic variables will include age, sex, race, ethnicity, height, weight, and body mass index (BMI). Baseline patient characteristics will include ASA status, physical examination findings, medical history, vital signs, clinical laboratory test results, and 12-lead ECG. Baseline patient characteristics will include prior medications.

## 7.4 Medical History

The number and percentage of patients with at least one medical history item in each System Organ Class (SOC) and preferred term will be presented overall and by treatment group, using the safety population.

Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

#### 8 EFFICACY ANALYSIS

## 8.1 Primary Efficacy

#### 8.1.1 Primary Efficacy Endpoint

The primary efficacy variable is success of the bronchoscopy procedure; a composite endpoint consisting of the following:

- Completion of the bronchoscopy procedure, AND
- No requirement for a rescue sedative medication, AND
- No requirement of more than 5 doses of study medication within any 15 minute window. For midazolam only: no requirement of more than 3 doses within any 12 minute window. (See section 6.2 for definition of how doses within a window are defined.)

Exceeding 5 doses within any sliding 15 minute window in the blinded (remimazolam or placebo) arm will be considered a treatment failure. Exceeding 3 doses within any 12 minute sliding window in the open-label midazolam arm will be considered a treatment failure.

#### 8.1.2 Primary Analysis

The primary efficacy analysis (success of the procedure using the composite endpoint) will be summarized descriptively for overall success for each treatment group, with summaries to include the number and percentage of patients.

Comparison of remimazolam and placebo

For the primary efficacy analysis, the following primary hypothesis will be tested:

H0: 
$$\pi_{\text{Remi}} \leq \pi_{\text{PLA}} \text{ vs. H1: } \pi_{\text{Remi}} > \pi_{\text{PLA}},$$

where  $\pi_{\text{Remi}}$  and  $\pi_{\text{PLA}}$  denote the success rates for Remimazolam and placebo, respectively. The primary efficacy analysis will be the comparison of these success rates between the remimazolam and placebo groups, using the Cochran-Mantel-Haenszel (CMH) test



Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017



The primary efficacy analysis will be based on the ITT, mITT and PP populations, with the mITT and PP population planned to confirm the results of the ITT population. *Comparison of remimazolam and midazolam* 

A 95% confidence interval of the comparison of success rates between midazolam and remimazolam will be presented but there will be no significance testing.



# 8.2 Secondary Efficacy

The following secondary efficacy variables will be presented with descriptive statistics by treatment group:

- 1. The **time to start of procedure** after administration of the first dose of randomized study medication.
- 2.
- 3. The **time to ready for discharge** (defined as ability to walk unassisted) after the end of bronchoscopy procedure (bronchoscope out).
- 4. The **time to ready for discharge** (defined as ability to walk unassisted) after the last injection of study drug.
- 5. The **time to fully alert** (time to first of three consecutive MOAA/S scores of 5) after the end of bronchoscopy procedure (bronchoscope out)).
- 6. The **time to fully alert** (time to first of three consecutive MOAAA/S scores of 5) after the last injection of study drug).

09 June 2017



All secondary efficacy variables will be compared between the three treatment groups. For the key secondary variables (variables 1-6), only the pairwise comparison between placebo and remimazolam will be used for exploratory efficacy significance testing. The time to event variables (variables 1-6, 13 above) will be analyzed by the logrank test. Kaplan-Meier graphs will also be fitted for each treatment group. Patients who do not reach fully alert will be censored at the time of their last MOAA/S assessment. Patients who do not reach ready for discharge criteria will be censored at the time of their last assessment. Median time to event with the corresponding 95% confidence interval will be presented. Additional quartiles (25% and 75%) and confidence intervals will be presented. A Cox's proportional hazard model including age group ( $<65, \ge 65$ ) will be fitted separately to the remimazolam and placebo, and the remimazolam and midazolam groups and the 95% confidence interval of the hazard ratio will be presented



Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

For the Readiness for Discharge score (variable 10) a value of 100 (= immediate readiness for discharge) will be used if the patient has already been discharged at the defined timepoint of analysis.



As a measure of discharge readiness, the proportion of the readiness for discharge score at 30, 60 and 90 minutes after t=0 will be compared across the treatment groups.

#### 9 SAFETY AND TOLERABILITY ANALYSIS

All safety analyses will be performed on the Safety Population, apart from the analyses of the Nellcor data which will use the Safety (Nellcor) populations.

All safety variables will be summarized descriptively. No statistical inference will be applied to the safety variables.

Safety variables that will be analyzed as safety endpoints include

- AEs, including adverse events with focus on respiratory and cardiovascular parameters and prolonged sedation (see <u>Appendix A</u>) and AEs potentially related to abuse (see <u>Appendix D</u>)
- Concomitant medication
- Clinical laboratory test results
- Vital signs (supine heart rate, systolic, diastolic and mean BP, respiration rate, temperature)
- Pulse oximetry measurements
- 12-lead and 3-lead ECG findings
- Physical examination finding



#### 9.1 Adverse Events

Treatment-emergent AEs (TEAEs) are defined as AEs reported at or after the start time of initial fentanyl administration or IMP, whatever is earlier, that are not present at Baseline, or that represent an exacerbation of an event that is present at Baseline. Any AE with an unknown start date and time will be considered treatment-emergent if the event does not discontinue prior to study drug administration.

The number and percentage of patients with TEAEs will be displayed for each treatment group by system organ class and preferred term using the current version of the Medical Dictionary for Regulatory Activities (MedDRA). Pretreatment AEs (reported from signing informed consent to before administration of study treatment) will be analyzed and displayed in a similar manner to TEAEs.

Summaries in terms of maximum severity and strongest relationship to study drug will also be provided.

Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

Summaries of serious adverse events (SAEs) similar to those of AEs will be provided separately. By-patient listings of AEs causing discontinuation of study drug and SAEs will be produced.

At each level of summarization (SOC or preferred term) a patient will be counted only once at the most severe or most related category. Patients with missing severity or relationship will be counted in the most severe and related category.

In addition, tachycardia (defined as heart rate recorded as >100 bpm, or an increase of 20% or more in the heart rate from baseline) will be analyzed.



The number and percentage of patients with AEs with a respiratory or cardiovascular focus will be displayed for each treatment group by system organ class (SOC) and preferred term, and also by standardised MedDRA query (SMQ) and preferred term. The preferred terms relating to these are shown in <u>Appendix A</u>.

The related AEs with a respiratory or cardiovascular focus will be displayed for each treatment group by system organ class and preferred term.

Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

The AEs with a respiratory or cardiovascular focus will be summarized split by time of onset (Day 1, after Day 1). The vital signs observed when a patient experienced a respiratory-cardiovascular AE will be summarized. The frequency of vital signs falling outside the normal range (as defined in the AE definitions above) will be given.

Interventions taken to prevent or treat these AEs are collected in the CRF. The number of patients requiring intervention and the type of interventions will be summarized.



# 9.2 Clinical Laboratory Tests

For qualitative clinical laboratory tests, the number and percentage of patients in each category will be displayed for each treatment group at each time point.

For all laboratory tests, a shift table will be produced summarizing changes from baseline to the end of the treatment period by treatment group.

Individual data listings of laboratory results will be presented for each patient at all study visits (scheduled and non-scheduled), including normal range limits for each laboratory test. Out-of-range results will be flagged, and determinations of whether the results were
09 June 2017

considered to be of clinical significance by the investigator will be included. Clinically significant laboratory test abnormalities that are considered AEs by the investigator will be presented in the AE summaries.

### 9.3 Vital Signs, Pulse Oximetry

Individual data listings of vital signs (supine heart rate, systolic and diastolic blood pressure, calculated mean arterial pressure, temperature, and respiration rate) will be presented for each patient at all visits (scheduled and non-scheduled). Pulse oximetry data (SpO<sub>2</sub>) will be presented by patient for pre-defined time points, and as the area under the oxygen desaturation curve (AUC<sub>Desat</sub>) over time from 1 minute before the first dose of randomized study drug to fully alert (AUC<sub>alert</sub>) and from 1 minute pre-dose to 20 minutes post dose (AUC<sub>20min</sub>). Desaturation is defined as an SpO<sub>2</sub> below 90%.

Descriptive statistics will be used to summarize the observed values at each time point, and the changes from baseline, for each treatment group. Graphic presentations of heart rate, blood pressure, and respiration rate may be presented by patients and as means by treatment over time. Vital sign and SpO<sub>2</sub> findings that were considered AEs by the Investigator will be presented by treatment in the AE summaries. The number of heart rate and SpO<sub>2</sub> findings (defined as being under the threshold value) that were not considered AEs as they did not meet the duration criteria will be presented by treatment, along with the duration.

The nadirs of heart rate, respiratory rate, and SpO<sub>2</sub>, after the first dose of randomized study drug of the data recorded in the CRF on the treatment day will be calculated and summarized by treatment group.

#### 9.3.1 Continuous Monitoring

The data from the Nellcor device used to perform continuous monitoring of heart rate, respiratory rate and SpO<sub>2</sub> (taken every second) during the procedure will be downloaded for analysis. All analyses of the Nellcor data will use the Safety (Nellcor) Populations.

The observational period will be from the first dose of any study medication (Fentanyl or IMP) until fully alert on the treatment day. Baseline will be defined as the pre-treatment values recorded in the CRF.

The nadirs and the peak for respiratory rate in the observational period will be identified and summarized by treatment group. If a "0" occurs then these values will be treated as missing data. Similarly, nadirs of heart rate and SpO<sub>2</sub> will be identified and summarized by treatment group.

All episodes of hypoxia (SpO2 <90%), bradycardia (heart rate <40 bpm), HR decreased (a drop in heart rate of 20% or more from baseline), respiratory depression (<8 breaths per minute) and respiratory increase (increase to >25 breaths per minute) in the observational period will be identified from the continuously recorded data. In addition, tachycardia (heart

09 June 2017

rate >100 bpm or increase of heart rate of 20% or more from baseline) will be analyzed. The number of patients reporting each type of AE and the duration will be summarized.

Further, those episodes of hypoxia, bradycardia or HR decreased which last long enough to match the protocol definitions of an AE above will be identified. The number of patients reporting episodes with a duration matching the AE definition and the number of patients with episodes with a duration that does not match the AE definition will be summarized, along with a summary of the durations of the episodes. Subgroup analyses of those AEs will be done as described in section 9.1.1 above.

The sites were asked whether they agreed that AEs identified in this way were actually AEs and whether they had been clinically observed and recorded in the CRF. The number of patients reporting each type of episode will be summarized by whether the investigator agreed.

#### 9.3.2 Continuous Monitoring – Exploratory Analyses

Further, exploratory analyses of the data collected with the Nellcor device may also be done after the main analyses of this study, and if so, those analyses will be described in a separate Exploratory SAP.

## 9.4 Electrocardiograms

#### 9.4.1 12-Lead ECG

The number and percentage of patients with normal and abnormal 12 lead ECG findings will be displayed for each treatment group at each time point. Additionally, patients with normal ECG findings at baseline and abnormal ECG findings at each time point will also be summarized by treatment group. For quantitative ECG variables (PR interval, RR interval, QRS interval, QT interval, and QT<sub>C</sub> interval [corrected using the Bazett and Fridericia formulae]), descriptive statistics will be given for the values themselves as well as for change from baseline, by treatment group at each time point.

#### 9.4.2 3-Lead ECG

The number and percentage of patients with normal and abnormal 3 lead ECG findings will be displayed for each treatment group at each time point. Additionally, patients with normal ECG findings at baseline and abnormal ECG findings at each time point will also be summarized by treatment group.

All episodes of bradycardia or other arrhythmias, captured in continuous 3-lead ECG recording, and any interventions that were instituted, will be documented and analyzed regardless of whether or not the event had been reported as an adverse event.

## 9.5 Physical Examinations

The number and percentage of patients with normal and abnormal physical examination findings will be displayed for each body system and treatment group at each time point.

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017

Additionally, patients with normal physical examination findings at baseline and abnormal physical examination findings at each time point will also be summarized by treatment group.



#### 9.7 Prior and Concomitant Medications

#### 9.7.1 Prior and Concomitant Medications

Prior and concomitant medication analyses will be provided for the safety population. Data on sedation rescue medication (which should only be midazolam) will be collected and presented separately from concomitant therapy as described in section 9.7.2.

All prior and concomitant medications will be coded using World Health Organization Drug Dictionary (WHO-DD) Version March 2015. Prior medications are defined as any medications taken prior to the start date of study treatment (whether stopped or continued after the start date of study treatment). Concomitant medications are defined as those used between the start date of study medication and the date of study completion or early termination. A medication could be flagged both as prior and concomitant if it was started prior to the patient's start date and continued on or after the start date of study medication.

Prior and concomitant medications will be summarized by treatment group in separate tables. Medications will be presented in alphabetical order, by Anatomical Therapeutic Class (ATC) (ATC Level 4) and preferred term. Tables will also show the overall number and percentage of patients receiving at least one medication. At each level of summarization (ATC class or preferred term) patients will be counted only once.

#### 9.7.2 Rescue Sedative Medications

The patient should receive midazolam as the rescue sedative at the discretion of the investigator, to allow for completion of the procedure or scope removal. The patient should also receive flumazenil as a reversal medication in case of remimazolam or midazolam overdose, or naloxone as a fentanyl antagonist. The number and percentage of patients receiving it will be summarized for all patients in the safety population by treatment group. A patient reporting rescue medication more than once will be counted once when calculating the number and percentage of patients.

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017



The number of patients where the number of doses of double-blind IMP was more than 5 within any 15 minute window or more than 3 doses within any 12 minute window in the midazolam arm will be considered a treatment failure, and will be calculated and summarized by treatment group.

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017



Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

## 11 REFERENCES

- 1. US Department of Health and Human Services. International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Rockville, MD: September 16, 1998. Federal Register;63(179):49583-49598..
- 2. ASA. (1999) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, August 7, 1999. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. The Royal Statistical Society: Code of Conduct, April 1993. http://www.rss.org.uk/main.asp?page=1875.

Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

# **12 ATTACHMENTS**

The table shells will be attached in a separate document.

09 June 2017

## APPENDIX A: Details of AEs with a Respiratory or Cardiovascular Focus

### LOW OXYGEN SATURATION/RESPIRATORY DEPRESSION

SMQ: Acute Central Respiratory Depression

#### Acute central respiratory depression (SMQ) [20000116]

| Name | Code | Level | Scope |
|-----------------------------------|----------|-------|--------|
| Acute respiratory failure | 10001053 | PT | Narrow |
| Apnoea | 10002974 | PT | Narrow |
| Apnoea neonatal | 10002976 | PT | Narrow |
| Apnoeic attack | 10002977 | PT | Narrow |
| Bradypnoea | 10006102 | PT | Narrow |
| Breath holding | 10006322 | PT | Narrow |
| Breath sounds abnormal | 10064780 | PT | Narrow |
| Breath sounds absent | 10062285 | PT | Narrow |
| Central-alveolar hypoventilation | 10007982 | PT | Narrow |
| Hypopnoea | 10021079 | PT | Narrow |
| Hypoventilation | 10021133 | PT | Narrow |
| Hypoventilation neonatal | 10021134 | PT | Narrow |
| Neonatal respiratory arrest | 10028968 | PT | Narrow |
| Neonatal respiratory depression | 10028970 | PT | Narrow |
| Neonatal respiratory failure | 10028975 | PT | Narrow |
| Postoperative respiratory failure | 10072651 | PT | Narrow |
| Respiratory arrest | 10038669 | PT | Narrow |
| Respiratory depression | 10038678 | PT | Narrow |

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017

### Acute central respiratory depression (SMQ) [20000116]

| Respiratory depth decreased | 10038681 | PT | Narrow |
|--------------------------------------------|----------|----|--------|
| Respiratory failure | 10038695 | PT | Narrow |
| Respiratory paralysis | 10038708 | PT | Narrow |
| Respiratory rate decreased | 10038710 | PT | Narrow |
| Alveolar oxygen partial pressure abnormal | 10068420 | PT | Broad |
| Alveolar oxygen partial pressure decreased | 10068419 | PT | Broad |
| Anoxia | 10002660 | PT | Broad |
| Apnoea test abnormal | 10074913 | PT | Broad |
| Asphyxia | 10003497 | PT | Broad |
| Bilevel positive airway pressure | 10064530 | PT | Broad |
| Blood gases abnormal | 10005539 | PT | Broad |
| Blood pH abnormal | 10005705 | PT | Broad |
| Blood pH decreased | 10005706 | PT | Broad |
| Capnogram abnormal | 10067661 | PT | Broad |
| Carbon dioxide abnormal | 10064156 | PT | Broad |
| Carbon dioxide increased | 10007225 | PT | Broad |
| Cardiac arrest | 10007515 | PT | Broad |
| Cardiac arrest neonatal | 10007516 | PT | Broad |
| Cardiopulmonary failure | 10051093 | PT | Broad |
| Cardio-respiratory arrest | 10007617 | PT | Broad |
| Cardio-respiratory arrest neonatal | 10007618 | PT | Broad |
| Cardio-respiratory distress | 10049874 | PT | Broad |
| Cheyne-Stokes respiration | 10008501 | PT | Broad |
| Continuous positive airway pressure | 10052934 | PT | Broad |
| Cyanosis | 10011703 | PT | Broad |

### Acute central respiratory depression (SMQ) [20000116]

| Cyanosis central | 10011704 | PT | Broad |
|----------------------------------------------------|----------|----|-------|
| Death neonatal | 10011912 | PT | Broad |
| Dependence on respirator | 10057482 | PT | Broad |
| Dyspnoea | 10013968 | PT | Broad |
| End-tidal CO2 abnormal | 10067663 | PT | Broad |
| End-tidal CO2 decreased | 10067665 | PT | Broad |
| Hyperbaric oxygen therapy | 10057480 | PT | Broad |
| Hypercapnia | 10020591 | PT | Broad |
| Hypercapnic coma | 10072597 | PT | Broad |
| Нурохіа | 10021143 | PT | Broad |
| Intermittent positive pressure breathing | 10052959 | PT | Broad |
| Life support | 10024447 | PT | Broad |
| Mechanical ventilation | 10067221 | PT | Broad |
| Mechanical ventilation complication | 10066821 | PT | Broad |
| Neonatal anoxia | 10028921 | PT | Broad |
| Neonatal asphyxia | 10028923 | PT | Broad |
| Neonatal hypoxia | 10050081 | PT | Broad |
| Neonatal respiratory acidosis | 10028966 | PT | Broad |
| Neonatal respiratory distress syndrome prophylaxis | 10054933 | PT | Broad |
| Oxygen saturation abnormal | 10033317 | PT | Broad |
| Oxygen saturation decreased | 10033318 | PT | Broad |
| Oxygen saturation immeasurable | 10051197 | PT | Broad |
| Oxygen supplementation | 10050322 | PT | Broad |
| PaO2/FIO2 ratio decreased | 10065413 | PT | Broad |
| PCO2 abnormal | 10058982 | PT | Broad |

09 June 2017

#### Acute central respiratory depression (SMQ) [20000116]

| PCO2 increased | 10034183 | PT | Broad |
|------------------------------------------|----------|----|-------|
| PO2 abnormal | 10062087 | PT | Broad |
| PO2 decreased | 10035768 | PT | Broad |
| Positive end-expiratory pressure | 10059890 | PT | Broad |
| Respiration abnormal | 10038647 | PT | Broad |
| Respiratory acidosis | 10038661 | PT | Broad |
| Respiratory disorder | 10038683 | PT | Broad |
| Respiratory disorder neonatal | 10061484 | PT | Broad |
| Respiratory distress | 10038687 | PT | Broad |
| Respiratory fume inhalation disorder | 10061485 | PT | Broad |
| Respiratory gas exchange disorder | 10062105 | PT | Broad |
| Respiratory therapy | 10059828 | PT | Broad |
| Sleep apnoea syndrome | 10040979 | PT | Broad |
| Venous oxygen partial pressure abnormal | 10068424 | PT | Broad |
| Venous oxygen partial pressure decreased | 10068423 | PT | Broad |
| Venous oxygen saturation abnormal | 10068428 | PT | Broad |
| Venous oxygen saturation decreased | 10068427 | PT | Broad |
| Ventilation perfusion mismatch | 10069675 | PT | Broad |
| Ventilation/perfusion scan abnormal | 10047265 | PT | Broad |
| Wean from ventilator | 10056353 | PT | Broad |
| Weaning failure | 10066829 | PT | Broad |

#### BRADYCARDIA:

Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017

- Bradyarrhythmias (incl conduction defects and disorders of sinus node function, SMQ):
  - Bradyarrhythmia
- Conduction defects (SMQ):

Atrial conduction time prolongation, Atrioventricular block, Atrioventricular block complete, Atrioventricular block first degree, Atrioventricular block second degree, atrioventricular dissociation, Bifascicular block, Bundle branch block, Bundle branch block bilateral, Bundle branch block left, Bundle branch block right, Conduction disorder, Defect conduction intraventricular, Electrocardiogram PQ interval prolonged, Electrocardiogram PR prolongation, Electrocardiogram QRS complex prolonged, Electrocardiogram QT prolonged, Long QT syndrome, Sinoatrial block, Trifascicular block, heart rate decreased

- Disorders of sinus node function (SMQ):

Sinus arrest, Sinus bradycardia, Sinus node dysfunction,

Should add: PT Bradycardia

#### HYPOTENSION:

• PTs: Blood pressure ambulatory decreased, blood pressure decreased, blood pressure diastolic decreased, blood pressure orthostatic decreased, blood pressure systolic decreased, mean arterial pressure decreased, pulmonary arterial pressure decreased, diastolic hypotension, hypotension, orthostatic hypotension, procedural hypotension, vasoplegia syndrome, orthostatic intolerance, presyncope, syncope

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017

#### HYPERTENSION:

## SMQ: Hypertension

## Hypertension (SMQ) [20000147]

| Name | Code | Level | Scope |
|----------------------------------------|----------|-------|--------|
| Accelerated hypertension | 10000358 | PT | Narrow |
| Blood pressure ambulatory increased | 10005732 | PT | Narrow |
| Blood pressure diastolic increased | 10005739 | PT | Narrow |
| Blood pressure inadequately controlled | 10051128 | PT | Narrow |
| Blood pressure increased | 10005750 | PT | Narrow |
| Blood pressure management | 10063926 | PT | Narrow |
| Blood pressure orthostatic increased | 10053355 | PT | Narrow |
| Blood pressure systolic increased | 10005760 | PT | Narrow |
| Diastolic hypertension | 10012758 | PT | Narrow |
| Eclampsia | 10014129 | PT | Narrow |
| Endocrine hypertension | 10057615 | PT | Narrow |
| Essential hypertension | 10015488 | PT | Narrow |
| Gestational hypertension | 10070538 | PT | Narrow |
| HELLP syndrome | 10049058 | PT | Narrow |
| Hyperaldosteronism | 10020571 | PT | Narrow |
| Hypertension | 10020772 | PT | Narrow |
| Hypertension neonatal | 10049781 | PT | Narrow |
| Hypertensive angiopathy | 10059238 | PT | Narrow |
| Hypertensive cardiomegaly | 10020801 | PT | Narrow |

| Protocol CNS7056-008 Statistical Analysis Plan | 09 June 2017 |
|------------------------------------------------|--------------|
|------------------------------------------------|--------------|

| Hypertensive cardiomyopathy | 10058222 | PT | Narrow |
|----------------------------------------|----------|----|--------|
| Hypertensive cerebrovascular disease | 10077000 | PT | Narrow |
| Hypertensive crisis | 10020802 | PT | Narrow |
| Hypertensive emergency | 10058179 | PT | Narrow |
| Hypertensive encephalopathy | 10020803 | PT | Narrow |
| Hypertensive heart disease | 10020823 | PT | Narrow |
| Hypertensive nephropathy | 10055171 | PT | Narrow |
| Labile hypertension | 10049079 | PT | Narrow |
| Malignant hypertension | 10025600 | PT | Narrow |
| Malignant hypertensive heart disease | 10025603 | PT | Narrow |
| Malignant renal hypertension | 10026674 | PT | Narrow |
| Maternal hypertension affecting foetus | 10026924 | PT | Narrow |
| Mean arterial pressure increased | 10026985 | PT | Narrow |
| Metabolic syndrome | 10052066 | PT | Narrow |
| Neurogenic hypertension | 10067598 | PT | Narrow |
| Orthostatic hypertension | 10065508 | PT | Narrow |
| Page kidney | 10076704 | PT | Narrow |
| Pre-eclampsia | 10036485 | PT | Narrow |
| Prehypertension | 10065918 | PT | Narrow |
| Procedural hypertension | 10062886 | PT | Narrow |
| Renal hypertension | 10038464 | PT | Narrow |
| Renal sympathetic nerve ablation | 10074864 | PT | Narrow |
| Renovascular hypertension | 10038562 | PT | Narrow |
| Retinopathy hypertensive | 10038926 | PT | Narrow |
| Secondary aldosteronism | 10039808 | PT | Narrow |

| Protocol CNS7056-008 Statistical Analysis Plan | 09 June 2017 |
|------------------------------------------------|--------------|
|------------------------------------------------|--------------|

# Hypertension (SMQ) [20000147]

| Secondary hypertension | 10039834 | PT | Narrow |
|-----------------------------------------|----------|----|--------|
| Systolic hypertension | 10042957 | PT | Narrow |
| Withdrawal hypertension | 10048007 | PT | Narrow |
| Aldosterone urine abnormal | 10061625 | PT | Broad |
| Aldosterone urine increased | 10001653 | PT | Broad |
| Angiotensin converting enzyme increased | 10049530 | PT | Broad |
| Angiotensin I increased | 10002488 | PT | Broad |
| Angiotensin II increased | 10002495 | PT | Broad |
| Blood aldosterone abnormal | 10005294 | PT | Broad |
| Blood aldosterone increased | 10005296 | PT | Broad |
| Blood catecholamines abnormal | 10005412 | PT | Broad |
| Blood catecholamines increased | 10005414 | PT | Broad |
| Blood pressure abnormal | 10005728 | PT | Broad |
| Blood pressure ambulatory abnormal | 10005730 | PT | Broad |
| Blood pressure diastolic abnormal | 10005736 | PT | Broad |
| Blood pressure fluctuation | 10005746 | PT | Broad |
| Blood pressure orthostatic abnormal | 10053354 | PT | Broad |
| Blood pressure systolic abnormal | 10005757 | PT | Broad |
| Catecholamines urine abnormal | 10061747 | PT | Broad |
| Catecholamines urine increased | 10061034 | PT | Broad |
| Diuretic therapy | 10053073 | PT | Broad |
| Ectopic aldosterone secretion | 10014148 | PT | Broad |
| Ectopic renin secretion | 10014171 | PT | Broad |
| Epinephrine abnormal | 10061845 | PT | Broad |
| Epinephrine increased | 10015064 | PT | Broad |

| Protocol CNS7056-008 Statistical Analysis Plan 09 . | June 2017 |
|-----------------------------------------------------|-----------|
|-----------------------------------------------------|-----------|

## Hypertension (SMQ) [20000147]

| Labile blood pressure | 10023533 | PT | Broad |
|-------------------------------------|----------|----|-------|
| Metanephrine urine abnormal | 10062193 | PT | Broad |
| Metanephrine urine increased | 10027445 | PT | Broad |
| Non-dipping | 10065226 | PT | Broad |
| Norepinephrine abnormal | 10061874 | PT | Broad |
| Norepinephrine increased | 10029752 | PT | Broad |
| Normetanephrine urine increased | 10049097 | PT | Broad |
| Pseudoaldosteronism | 10037113 | PT | Broad |
| Renin abnormal | 10038556 | PT | Broad |
| Renin increased | 10038559 | PT | Broad |
| Renin-angiotensin system inhibition | 10049415 | PT | Broad |
| Tyramine reaction | 10067895 | PT | Broad |

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017

#### PROLONGED SEDATION

SMQ: Anticholinergic Syndrome plus single PTs

## Anticholinergic syndrome (SMQ) [20000048]

| Name | Code | Level | Scope |
|------------------------------------|----------|-------|--------|
| Anticholinergic syndrome | 10002757 | PT | Narrow |
| Ataxia | 10003591 | PT | Broad |
| Autonomic nervous system imbalance | 10003840 | PT | Broad |
| Balance disorder | 10049848 | PT | Broad |
| Coordination abnormal | 10010947 | PT | Broad |
| Depressed level of consciousness | 10012373 | PT | Broad |
| Dizziness | 10013573 | PT | Broad |
| Hyporesponsive to stimuli | 10071552 | PT | Broad |
| Loss of consciousness | 10024855 | PT | Broad |
| Presyncope | 10036653 | PT | Broad |
| Sedation | 10039897 | PT | Broad |
| Slow response to stimuli | 10041045 | PT | Broad |
| Somnolence | 10041349 | PT | Broad |
| Stupor | 10042264 | PT | Broad |
| Agitation | 10001497 | PT | Broad |
| Confusional state | 10010305 | PT | Broad |
| Delirium | 10012218 | PT | Broad |
| Disorientation | 10013395 | PT | Broad |
| Hallucination | 10019063 | PT | Broad |

| Protocol CNS7056-008 Statistical Analysis Plan | 09 June 2017 |
|------------------------------------------------|--------------|
|------------------------------------------------|--------------|

| Anticholinergic syndrome (SMQ) [20000048] |
|-------------------------------------------|

| Hallucination, auditory | 10019070 | PT | Broad |
|-----------------------------|----------|----|-------|
| Hallucination, gustatory | 10019071 | PT | Broad |
| Hallucination, olfactory | 10019072 | PT | Broad |
| Hallucination, synaesthetic | 10062824 | PT | Broad |
| Hallucination, tactile | 10019074 | PT | Broad |
| Hallucination, visual | 10019075 | PT | Broad |
| Hallucinations, mixed | 10019079 | PT | Broad |
| Restlessness | 10038743 | PT | Broad |
| Thinking abnormal | 10043431 | PT | Broad |
| Abasia | 10049460 | PT | Broad |
| Accommodation disorder | 10000389 | PT | Broad |
| Anhidrosis | 10002512 | PT | Broad |
| Blindness transient | 10005184 | PT | Broad |
| Cycloplegia | 10011719 | PT | Broad |
| Dry eye | 10013774 | PT | Broad |
| Dry mouth | 10013781 | PT | Broad |
| Dysphagia | 10013950 | PT | Broad |
| Gait disturbance | 10017577 | PT | Broad |
| Hemifacial anhidrosis | 10075470 | PT | Broad |
| Hyperaemia | 10020565 | PT | Broad |
| Hyperpyrexia | 10020741 | PT | Broad |
| Hypohidrosis | 10021013 | PT | Broad |
| Mydriasis | 10028521 | PT | Broad |
| Pyrexia | 10037660 | PT | Broad |
| Tachycardia | 10043071 | PT | Broad |

Protocol CNS7056-008 Statistical Analysis Plan 09 June 2017

### Anticholinergic syndrome (SMQ) [20000048]

| Thirst | 10043458 | PT | Broad |
|-----------------------------------|----------|----|-------|
| Toxicity to various agents | 10070863 | PT | Broad |
| Urinary retention | 10046555 | PT | Broad |
| Vision blurred | 10047513 | PT | Broad |
| Visual acuity reduced | 10047531 | PT | Broad |
| Visual acuity reduced transiently | 10047532 | PT | Broad |

Add PTs: Sedation, Post-injection delirium sedation syndrome, Reversal of sedation

09 June 2017

## **APPENDIX B: Diseases of Interest for Drug-Disease Interaction Analysis**

| Disease | Preferred Terms |
|---|---|
| Congestive Heart Failure | Cardiac failure (SMQ) |
| Arterial Hypertension | Hypertension (SMQ) |
| Coronary artery disease | Ischaemic heart disease (SMQ), including both Myocardial infarction (SMQ) and Other ischaemic heart disease (SMQ) In addition other coronary artery diseases, not related with ischaemic heart disease include: Arteritis coronary, Coronary artery aneurysm, Coronary artery perforation, Coronary artery dilatation, Coronary artery stent removal, Chest discomfort, and Chest pain. |
| Chronic obstructive pulmonary disease | Chronic obstructive pulmonary disease,<br>Bronchitis chronic, Infective exacerbation<br>of chronic obstructive airways disease,<br>asthma. |
| Pre-existing mental impairment (e.g. dementia) | Mental disability, Mental retardation, Mild mental retardation, Moderate mental retardation, Profound mental retardation, Severe mental retardation, Mental status changes postoperative, Mental disorder due to a general medical condition. Dementia (SMQ) |
| | Psychosis and psychotic disorders (SMQ) |
| Gastrointestinal disorder | GI non-specific inflammation and dysfunctional conditions (SMQ) and GI perforation, ulceration, haemorrhage or obstruction (SMQ) |



| • <u> </u> |
|------------|
| 1 |
| • |
| ' |

Protocol CNS7056-008 Statistical Analysis Plan

09 June 2017



09 June 2017



09 June 2017



